CLINICAL TRIAL: NCT02907307
Title: Comparative Study of the Efficacy and Safety of LactiSal 1% Vaginal Gel and LactSal 50 mg Vaginal Tablet Versus Clotrimazole 100 mg Vaginal Tablet in the Treatment of Vulvovaginal Candidiasis (VVC)
Brief Title: Efficacy, Safety LactiSal 1% Gel, LactSal 50 mg, Clotrimazole 100 mg Tablet in Treatment Vulvovaginal Candidiasis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Development project stopped
Sponsor: Medinova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LacS011
Record Dates: First submitted 2015-09-23; First posted 2016-09-20 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2017-12

CONDITIONS: Vulvovaginal Candidiasis
Keywords: LactiSal; Vaginal therapy
MeSH Terms: conditions — Candidiasis, Vulvovaginal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LactiSal vaginal gel 1% (Experimental): 5g of 1%LactiSal Gel vaginal gel once daily for 6 days
  Interventions: Device: LactiSal vaginal gel 1%
- LactiSal vaginal tablet 50 mg (Experimental): 50 mg of LactiSal vaginal tablet daily for 6 days
  Interventions: Device: LactiSal vaginal tablet 50mg
- Clotrimazole vaginal tablet 100mg (Active Comparator): 100 mg Clotrimazole vaginal tablet daily for 6 days
  Interventions: Drug: Clotrimazole vaginal tablet 100mg

INTERVENTIONS:
Device: LactiSal vaginal gel 1% — to be administered daily intravaginally for 6 days
  Arms: LactiSal vaginal gel 1%
Device: LactiSal vaginal tablet 50mg — to be administered daily intravaginally for 6 days
  Arms: LactiSal vaginal tablet 50 mg
Drug: Clotrimazole vaginal tablet 100mg — to be administered daily intravaginally for 6 days
  Other Names: Candibene
  Arms: Clotrimazole vaginal tablet 100mg

SUMMARY:
The purpose of this study is to compare the efficacy and safety of LactiSal 1%vaginal gel and LactiSal 50 mg vaginal tablet with the standart treatment of clotrimazole 100 mg vaginal tablet in woman with vulvovaginal candidiasis (VVC)

DETAILED DESCRIPTION:
National multicenter,randomized, open-label, active-controlled with three parallel groups.Eligible patients are randomized to receive LactiSal 1% vaginal gel, LactiSal 50 mg vaginal tablet or clotrimazole 100 mg vaginal tablet for 6 days. Control examaminations are performed 10 after entry and 4 weeks after control visit 1.

The study investigates the clinical efficacy and safety of Lactisal 1% vaginal gel and LactiSal 50mg vaginal tablets in the intended use, i.e. vaginal application, and the following intended claims:

* Treatment of vaginal yeast vaginitis
* Relieves vaginal itching, burning, redness and discharge in case of yeast vaginitis
* Inhibition of yeast colonization in the vagina in case of yeast vaginitis. The study is designed to compare the clinical efficacy and safety of Lactisal 1% vaginal gel and LactiSal 50 mg vaginal tablets to a current standard drug therapy, i.e. clotrimazole 100 mg vaginal tablets.

While LactiSal is classified as medical device class IIa, the comparator is a medicinal (pharmaceutical) product. The study represents a "mixed" study, comparing the efficacy of a medical device with a pharmaceutical product.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical signs & symptoms of VVC as Total Severity Score, TSC 4 (range 0-15):

   * vaginal itching (range 0-3) ,
   * vaginal burning or soreness (range 0-3),
   * abnormal vaginal discharge (range 0-3),
   * vulvo/vaginal erythema or oedema (range 0-3),
   * vulvar excoriation or fissure formation (range 0-3).
2. Direct microscopy (Wet smear) positive for yeast forms (hyphae, pseudohyphae) or budding yeasts
3. Normal vaginal pH (≤4.5)
4. Age: 18 years and older
5. Signed Written Informed Consent to participate in this study.

Exclusion Criteria:

* Recurrent VVC (4 episodes of VVC in the past 12 months).
* Women with other vaginal infections, e.g. bacterial vaginosis, aerobic vaginitis, trichomoniasis, and mixed infections.
* Women using oral or vaginal antifungals within 2 weeks prior to enrolment.
* Women using any intra-vaginal products, also vaginal douches containing soaps and other anionic, surface-active substances, within 2 weeks prior to enrolment.
* Women using any antibiotic or anti-infective within 2 weeks prior to enrolment.
* Women having menstruation bleeding at enrolment
* Cervicitis, cervical erosions, and malignant tumours in the genital tract
* Pregnancy or lactation.
* Women not consenting to be sexually abstinent during the treatment, not taking oral contraceptive or not having an IUD for contraception
* Woman using intravaginal pessaries, rings, sponges or diaphragms
* Severe systemic diseases (diabetes mellitus, cancer, tuberculosis, autoimmune diseases, severe psychiatric conditions, etc.).
* Women with confirmed or suspected STD (HIV infection, gonorrhoea, syphilis, chlamydiasis, etc.).
* Known or suspected hypersensitivity to one of the study medications, inclusive their excipients.
* Participation of patient in another clinical study concomitantly or within 30 days prior to enrolment
* Patient is relative of, or staff directly reporting to, the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate | 10 days after entry (C1)
  Clinical cure is defined as patient having a Total Severity Score of less than 3. The Total Severity Score (TSC) is assessed by the Investigator, examining and interviewing the patient. The TSC is the sum score of the 5 individual signs symptoms - vaginal itching, vaginal burning or soreness, abnormal vaginal discharge, vulvovaginal erythema or oedema and vulval excoriation or fissure formation. Each sign and symptom is assessed with a score from 0 to 3, resulting in total score for TSC of 0 to 15.

SECONDARY OUTCOMES:
Clinical cure rate | 4 weeks after control visit 1
  Clinical cure is defined as patient having a Total Severity Score of less than 3. The Total Severity Score (TSC) is assessed by the Investigator, examining and interviewing the patient. The TSC is the sum score of the 5 individual signs symptoms - vaginal itching, vaginal burning or soreness, abnormal vaginal discharge, vulvovaginal erythema or oedema and vulval excoriation or fissure formation. Each sign and symptom is assessed with a score from 0 to 3, resulting in total score for TSC of 0 to 15.
Microbiological cure rate | 10 days after entry visit and 4 weeks after control visit 1
  Negative for Candida in microscopy and culture
Therapeutic cure rate | 10 days after entry visit and 4 weeks after control visit 1
  Clinically and microbiologically cure combined
The Total Severity Score (TSC) Individual clinical signs and symptoms | 10 days after entry visit and 4 weeks after control visit 1
  The TCS assessed by the investigator
  * vaginal itching (range 0-3)
  * vaginal burning or soreness (range 0-3)
  * abnormal vaginal discharge (range 0-3)
  * vulvo/vaginal erythema or oedema (range 0-3)
  * vulvar excoriation or fissure formation (range 0-3)
Dyspareunia and external dysuria | 10 days after entry visit and 4 weeks after control visit 1
  Presence of dyspareunia and external dysuria (yes/no)
Direct microscopy (Wet smear) | 10 days after entry visit and 4 weeks after control visit 1
  Number of positive findings in Direct microscopy (Wet smear) in comparison to visit E
pH | 10 days after entry visit and 4 weeks after control visit 1
  Mean vaginal pH in comparison to visit E
Candida culture | 10 days after entry visit and 4 weeks after control visit 1
  Number of positive Candida cultures in comparison to visit E
Efficacy assessment | 10 days after entry visit and 4 weeks after control visit 1
  Global assessment of efficacy by patient and investigator
Patients diary | 10 days after entry visit and 4 weeks after control visit 1
  Assessment clinical symptoms from patient?s diary
Patient's satisfaction | 10 days after entry visit and 4 weeks after control visit 1
  Patient will be asked how satisfied she was with the treatment received based on 8 standardized questions.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Halaška, MD, Principal Investigator — Nemocnice Bulovka, 1. LF UK

IPD SHARING:
Plan to Share IPD: Undecided